CLINICAL TRIAL: NCT00416000
Title: Phase 1 Study of Complement Activation Following Ruptured Abdominal Aortic Aneurysm: Combining Human Observation With Animal Experimentation to Establish a Framework for Human Therapy
Brief Title: Mechanism and Prevention of Remote Organ Injury Following Ruptured Aortic Aneurysm
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Thomas Lindsay, Professor of Surgery, University Health Network, Toronto
Other Study IDs: 06-0671B
Record Dates: First submitted 2006-12-22; First posted 2006-12-27 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Open/Elective EVAR patients
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
It has been estimated that 80% of deaths from abdominal aortic aneurysms results from rupture. Endovascular Aneurysm Repair (EVAR) has been applied to RAAA (Ruptured Abdominal Aortic Aneurysm) patients with reports of improvements. Despite the use of EVAR, patients have developed complications with lung and kidney function. This study will investigate certain biochemical processes that will potentially reduce these complications. Knowledge gained from this study may also be used to further research in this field through larger studies.

ELIGIBILITY:
Inclusion Criteria:

* Open/Elective EVAR patients

Exclusion Criteria:

* Patients who do not present with abdominal aortic aneurysms or ruptured abdominal aortic aneurysm

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those undergoing AAA repair for elevtive and ruptured AAA by both EVAR and open methods.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days

SECONDARY OUTCOMES:
multiple organ failure | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Lindsay, MD, Principal Investigator — TGH, UHN
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada